CLINICAL TRIAL: NCT05290805
Title: Optimized CT-imaging Protocol in VA-ECMO Patients After Cardiopulmonary Resuscitation - a Single-center Prospective Non-randomized Cohort Study
Brief Title: Optimized CT-imaging Protocol in VA-ECMO Patients After CPR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Philipp Dominik Stelzer, Principal Investigator, MD, Medical University of Vienna
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: EK-Nr. 1941/2021
Record Dates: First submitted 2022-02-21; First posted 2022-03-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Cardiopulmonary Arrest; VA-ECMO
Keywords: CPR; ECMO; Vessel opacification; Computed tomography
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ECMO flow rate reduction (Experimental): In the intervention cohort ECMO flow rate is reduced for the duration of CT image acquisition (max. 1-2 min.), if the hemodynamic and respiratory situation allows it. Feasibility is determined by the accompanying emergency physician right before the CT scan and adapted to the individually tolerable level (max. 50% of initial flow, no less than 1,5 litre/min). After image acquisition, ECMO flow rate is immediately returned to the initial or clinically optimal value at this moment.
  Interventions: Diagnostic Test: ECMO flow rate reduction
- no ECMO flow rate reduction (No Intervention): In this cohort ECMO flow rate is not reduced for CT image acquisition.

INTERVENTIONS:
Diagnostic Test: ECMO flow rate reduction — ECMO flow rate is reduced for the duration of CT image acquisition (max. 1-2 min.), if the hemodynamic and respiratory situation allows it. Feasibility is determined by the accompanying emergency physician right before the CT scan and adapted to the individually tolerable level (max. 50% of initial flow, no less than 1,5 litre/min). After image acquisition, ECMO flow rate is immediately returned to the initial or clinically optimal value at this moment.
  Arms: ECMO flow rate reduction

SUMMARY:
Veno-arterial (VA) extracorporal membrane oxygenation (ECMO) is an increasingly applied method in patients under cardiopulmonary resuscitation (CPR), who are regularly examined with a contrast-enhanced computed tomography to search for the underlying pathology as well as complications from the implantation of the ECMO system or CPR. The extraordinary hemodynamic situation due to VA-cannulation with antegrade and retrograde perfusion is a challenge to the diagnostically required simultaneous opacification of pulmonary and systemic arterial vessels. Evidence regarding the effect of ECMO flow rate, cannula position, cardiac function and contrast agent injection site is scarce and to the best of the authors' knowledge, no standardized scan protocol for this patient collective exists.

In this study, all adult emergency department patients at our institution with femoro-femoral VA-ECMO and ongoing or recent cardiopulmonary resuscitation, who are referred to a clinically indicated CT scan in this context, will be included, aiming for a total of n=50 patients. The first 25 consecutive patients will be assigned to the intervention cohort. For these patients the ECMO flow rate is reduced by a maximum of 50% of initial flow, but to no less than 1,5 liter/min, for the duration of the CT scan (max. 1-2 minutes), given the hemodynamic and respiratory situation allows it. The following 25 consecutive patients will be assigned to the control cohort for whom ECMO flow rate is not reduced. Clinical data (e.g. ECMO flow rate, ventilation parameters, cardiac function, venous line for contrast injection) at the time of imaging will be documented via a standardized data sheet. The applied CT protocol routinely comprises a non-contrast-enhanced cranial CT (CCT), CT angiography (CTA) of the aorta as well as a portal-venous phase of the chest and abdomen. Complementary scans will be performed as clinically indicated.

The aim of this single-center prospective cohort study is to evaluate the performance of an optimized CT protocol for this patient cohort and whether a reduction of ECMO flow rate improves contrast enhancement of critically relevant vessels in these CT examinations in comparison to a non-reduction cohort.

DETAILED DESCRIPTION:
Background:

Extracorporal membrane oxygenation (ECMO) is an increasingly applied method of last resort for treating severe respiratory or combined cardiopulmonary failure. Different configurations of cannulation, either veno-venous (VV) or veno-arterial (VA), are used depending on indication. The latter is commonly used in patients under cardiopulmonary resuscitation to temporarily provide adequate organ-perfusion until the underlying pathology is found and treated. Alas being a revolutionary method, there is also a non-negligible number of vascular complications due to necessary insertion of cannulas in large vessels in combination with full anticoagulation. Therefore, these patients are regularly examined with a subsequent contrast-enhanced computed tomography to rule out complications and search for potential underlying causes of cardiac arrest. However, the extraordinary hemodynamic situation resulting from VA-cannulation with antegrade and retrograde perfusion challenges the diagnostically required simultaneous opacification of pulmonary and systemic arterial vessels. In this setting, siphoning, mixing and dilution effects of contrast agent and non-contrasted blood often cause incomplete or inhomogeneous vessel contrast, rendering exams partially non-diagnostic. Evidence regarding the effect of cannula position, ECMO flow rate, cardiac function and contrast agent injection site is scarce and as yet, to the best of the authors' knowledge, no standardized scan protocol for this patient collective exists.

Methods:

All adult emergency department patients at the Vienna General Hospital with femoro-femoral VA-ECMO and undergoing or recent cardiopulmonary resuscitation, who are subsequently referred to a clinically indicated CT scan for the detection of causes and complications or their exclusion, will be included in this study, aiming for a total of n=50 patients. The first 25 consecutive patients will be assigned to the intervention (flow reduction) cohort and the following 25 consecutive patients will be assigned to the control (no flow reduction) cohort. Clinical data (e.g. ECMO flow rate, ventilation parameters, cardiac function, venous line for contrast injection) at the time of imaging will be retrieved from the accompanying treating physician and are documented via a standardized data sheet.

In the intervention cohort ECMO flow rate is reduced for the duration of contrast administration and acquisition of an arterial and venous phase of the whole body (max. 1-2 minutes) given the hemodynamic and respiratory situation allows it. Whether this is possible, is determined right before the CT scan by the accompanying emergency physician and adapted to the individually tolerable level (max. 50% of initial flow, no less than 1,5 liter/min). After image acquisition, ECMO flow rate is then immediately returned to the initial or clinically optimal value at this moment. If the patient shows any signs of instability during this short period of imaging acquisition, the scan will be interrupted and immediate countermeasures will be taken by the accompanying team of emergency physicians and nurses. During the examination the vital signs of all patients are permanently monitored. The applied CT protocol is the established protocol at our department and comprises a non-contrast-enhanced cranial CT (CCT), CT angiography (CTA) of the aorta as well as a portal-venous phase of the chest and abdomen. Complementary scans, e.g. CT of cervical spine or CTA of cerebral arteries, will be performed as clinically indicated. After the examination, ECMO flow rate will be increased to the initial or at this point clinically optimal value and the acquired images are, within clinical routine, immediately reviewed and reported by the radiologist in charge. Diagnostic quality of the acquired images, vessel opacification, the impact of CT findings and diagnoses on clinical management as well as resulting management changes will be documented and analyzed.

Aims:

The aim of this single-center prospective cohort study is to evaluate the performance of an optimized CT protocol and whether a reduction of ECMO flow rate improves contrast enhancement of critically relevant vessels in CT examinations of patients after cardiopulmonary resuscitation with femoro-femoral VA-ECMO (eCPR) in comparison to a non-reduction cohort.

ELIGIBILITY:
Inclusion Criteria:

* Running or recent eCPR
* Clinically indicated CT and CT angiography of chest and abdomen (and head, if required)
* Femoro-femoral VA-ECMO-cannulation

Exclusion Criteria:

- Contraindication for CT scan or administration of iodinated contrast agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Computed tomography vessel opacification | Three years
  To assess and compare overall vessel opacification of eCPR patients with and without ECMO flow reduction, measured by mean HU in a representative cross-section of clinically relevant vessels.
Number and clinical impact of pathological findings | ten days
  To assess the number and clinical impact of additional / previously unknown pathological findings in eCPR patients detected by early post-eCPR CT, measured by direct feedback of the treating emergency physician on the relevance (Likert scale 1-5) and consequences (time and type) of findings.

SECONDARY OUTCOMES:
Subjective CT image quality | Three years
  To assess whether flow reduction improves subjective CT image quality compared to the no-flow reduction cohort, measured by a Likert-Scale from 1-5.
CT vessel opacification homogeneity | Three years
  To assess whether flow reduction results in a more homogeneous vessel opacification, measured by standard deviation of HU in a representative cross-section of clinically relevant vessels.
Follow-up CT exams | Three years
  To assess whether an all-in-one exam before ICU admission reduces number of follow-up CT exams, radiation dose and/or contrast agent dose, measured by comparing cumulative exam numbers, radiation and contrast agent dose of the study cohort to a retrospective cohort of eCPR exams.
Correlations between mean vessel opacification, subjective image quality and appearance of artifacts with intrinsic and extrinsic factors | Three years
  To find correlations between intrinsic and extrinsic factors and mean vessel opacification, subjective image quality and appearance of artifacts, measured by correlation of mean HU for metric variables and uni- and multivariate analysis for binary variables.

CONTACTS AND LOCATIONS:
Overall Officials: Dietmar Tamandl, MD, Assoc.-Prof., Study Director — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lambert L, Grus T, Balik M, Fichtl J, Kavan J, Belohlavek J. Hemodynamic changes in patients with extracorporeal membrane oxygenation (ECMO) demonstrated by contrast-enhanced CT examinations - implications for image acquisition technique. Perfusion. 2017 Apr;32(3):220-225. doi: 10.1177/0267659116677308. Epub 2016 Oct 31. PMID 27799498
- [Background] Auzinger G, Best T, Vercueil A, Willars C, Wendon JA, Desai SR. Computed tomographic imaging in peripheral VA-ECMO: where has all the contrast gone? J Cardiothorac Vasc Anesth. 2014 Oct;28(5):1307-9. doi: 10.1053/j.jvca.2013.06.027. Epub 2013 Oct 30. No abstract available. PMID 24183316
- [Background] Kohler K, Valchanov K, Nias G, Vuylsteke A. ECMO cannula review. Perfusion. 2013 Mar;28(2):114-24. doi: 10.1177/0267659112468014. Epub 2012 Dec 20. PMID 23257678
- [Background] Lee S, Chaturvedi A. Imaging adults on extracorporeal membrane oxygenation (ECMO). Insights Imaging. 2014 Dec;5(6):731-42. doi: 10.1007/s13244-014-0357-x. Epub 2014 Oct 9. PMID 25296619
- [Background] Acharya J, Rajamohan AG, Skalski MR, Law M, Kim P, Gibbs W. CT Angiography of the Head in Extracorporeal Membrane Oxygenation. AJNR Am J Neuroradiol. 2017 Apr;38(4):773-776. doi: 10.3174/ajnr.A5060. Epub 2017 Jan 5. PMID 28057636
- [Background] Gullberg Lidegran M, Gordon Murkes L, Andersson Lindholm J, Frenckner B. Optimizing Contrast-Enhanced Thoracoabdominal CT in Patients During Extracorporeal Membrane Oxygenation. Acad Radiol. 2021 Jan;28(1):58-67. doi: 10.1016/j.acra.2020.01.029. Epub 2020 Feb 21. PMID 32094031
- [Background] Yang KJ, Wang CH, Huang YC, Tseng LJ, Chen YS, Yu HY. Clinical experience of whole-body computed tomography as the initial evaluation tool after extracorporeal cardiopulmonary resuscitation in patients of out-of-hospital cardiac arrest. Scand J Trauma Resusc Emerg Med. 2020 Jun 11;28(1):54. doi: 10.1186/s13049-020-00746-5. PMID 32527321
- [Background] Zotzmann V, Rilinger J, Lang CN, Duerschmied D, Benk C, Bode C, Wengenmayer T, Staudacher DL. Early full-body computed tomography in patients after extracorporeal cardiopulmonary resuscitation (eCPR). Resuscitation. 2020 Jan 1;146:149-154. doi: 10.1016/j.resuscitation.2019.11.024. Epub 2019 Dec 4. PMID 31811881
- [Background] Holmberg MJ, Geri G, Wiberg S, Guerguerian AM, Donnino MW, Nolan JP, Deakin CD, Andersen LW; International Liaison Committee on Resuscitation's (ILCOR) Advanced Life Support and Pediatric Task Forces. Extracorporeal cardiopulmonary resuscitation for cardiac arrest: A systematic review. Resuscitation. 2018 Oct;131:91-100. doi: 10.1016/j.resuscitation.2018.07.029. Epub 2018 Jul 29. PMID 30063963